CLINICAL TRIAL: NCT04976595
Title: A 24-hour Ambulatory Blood Pressure Monitoring Study in Hypogonadal Men Treated With Natesto Nasal Testosterone Gel
Brief Title: A Study to Monitor Ambulatory Blood Pressure Monitoring in Hypogonadal Men Treated With Nasal Testosterone Gel
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acerus Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAT-2020-01
Record Dates: First submitted 2021-07-16; First posted 2021-07-26 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Hypogonadism
Keywords: Hypogonadism; Gonadal Disorders; Testosterone; Hormones; Androgens; Endocrine System Diseases; Ambulatory Blood Pressure Monitoring
MeSH Terms: conditions — Hypogonadism; Gonadal Disorders; Endocrine System Diseases | interventions — Natesto

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Natesto (Experimental): Participants will administer Natesto, gel, intranasally, three times daily up to Day 120. A multiple-dose dispenser will be used for gel deposition into the nasal cavity.
  Interventions: Drug: Natesto

INTERVENTIONS:
Drug: Natesto — Nasal gel containing testosterone 11 mg/dose (5.5 mg/nostril) three times daily.
  Other Names: Testosterone Nasal Gel

SUMMARY:
The purpose of this study is to assess the change in 24-hour ambulatory blood pressure monitoring (ABPM) between baseline (Day 0) and Day 120 following 4 months of testosterone therapy with Natesto.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign and date the study consent form(s) which have been approved by an Institutional Review Board (IRB). Written consent must be obtained prior to the initiation of any study procedures.
* Male between 18 and 80 years of age, inclusive, with documented onset of hypogonadism prior to age 65.
* Serum total testosterone < 300 ng/dL based on 2 consecutive blood samples obtained no greater than 1-4 weeks apart between 6 and 10 AM following an appropriate washout of current androgen replacement therapy if not testosterone naive. Historical values from the past 6 months may be used.
* Testosterone Therapy naive, OR off any testosterone therapy for at least 4 months OR agree to a 4-month washout of current testosterone therapy prior to entry at Visit 1.
* Average office blood pressure measurement <140 millimetre of mercury (mmHg) SBP -AND- <90 mmHg DBP.
* If the participant is on an antihypertensive regimen, he has been on it for at least 4 weeks.
* Judged to be in good general health as determined by the principal investigator based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* History of significant sensitivity or allergy to androgens, castor oil or product excipients.
* Clinically significant findings in the pre-study examinations including abnormal breast examination requiring follow-up, an abnormal ECG.
* Abnormal prostate digital rectal examination (DRE) with palpable nodule(s) or International Prostate Symptom Score (I-PSS) score > 19 points.
* Body mass index (BMI) ≥ 35 kg/m^2.
* Clinically significant abnormal laboratory value, in the opinion of the investigator, in serum chemistry, hematology, or urinalysis including but not limited to:

  * Prostate specific antigen (PSA) > 4 ng/mL
  * Hematocrit < 35% or > 50%
  * Baseline hemoglobin > 16 g/dL
  * Hemoglobin A1C (HbA1C) > 9.0%
  * Estimated glomerular filtration rate (eGFR) <45
* History of seizures or convulsions, including febrile, alcohol or drug withdrawal seizures.
* History of any clinically significant illness, infection, or surgical procedure within 4 weeks prior to study drug administration except for diabetes, or renal disease.
* History of stroke or myocardial infarction within the past 5 years.
* History of, or current or suspected, prostate or breast cancer.
* History of diagnosed, severe, untreated, obstructive sleep apnea.
* History of abuse of alcohol or any drug substance in the opinion of the investigator within the previous 2 years.
* Currently using tobacco, e-cigarettes or other nicotine containing products.
* History of nasal disorders such as nasal surgery; nasal trauma resulting in nasal fracture within the previous 6 months or nasal fracture that caused a deviated anterior nasal septum; or sinus surgery or sinus disease.
* Receipt of any investigational product within 4 weeks of study start.
* Inability to understand and provide written informed consent for the study.
* Considered by the investigator or the sponsor-designated physician, for any reason, as an unsuitable candidate to receive Natesto.
* Participants working night-shifts.
* Participants performing strenuous manual labor while wearing the ABPM monitor.
* Participants with chronic atrial fibrillation (interferes with the ability to obtain precise ambulatory recordings).

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 218 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in 24-Hour Systolic Blood Pressure (SBP) At Day 120 | Baseline (Day 0) and Day 120
  The change from baseline (Day 0) in 24-hour SBP after 120 days of Natesto treatment will be assessed.

SECONDARY OUTCOMES:
Change From Baseline in 24-hour Average Mean Arterial Pressure (MAP) | Baseline (Day 0) up to Day 120
Change From Baseline in 24-hour Average Systolic Blood Pressure (SBP) | Baseline (Day 0) up to Day 120
Change From Baseline in 24-hour Average Diastolic Blood Pressure (DBP) | Baseline (Day 0) up to Day 120
Change From Baseline in 24-hour Average Pulse Pressure | Baseline (Day 0) up to Day 120
Change From Baseline in 24-hour Average Heart Rate | Baseline (Day 0) up to Day 120
Change From Baseline in Hourly Average Mean Arterial Pressure (MAP) | Baseline (Day 0) up to Day 120
Change From Baseline in Hourly Average Systolic Blood Pressure (SBP) | Baseline (Day 0) up to Day 120
Change From Baseline in Hourly Average Diastolic Blood Pressure (DBP) | Baseline (Day 0) up to Day 120
Change From Baseline in Hourly Average Pulse Pressure | Baseline (Day 0) up to Day 120
Change From Baseline in Hourly Average Heart Rate | Baseline (Day 0) up to Day 120
Percentage of Participants With New Anti-hypertensive Medications | Baseline (Day 0) up to Day 120
Percentage of Participants With Dose Increases in Anti-hypertensive Medications | Baseline (Day 0) up to Day 120

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Horizon Clinical Research Associates, Phoenix, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - Valley Clinical Trials, Northridge, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Florida Healthcare Associates, Boynton Beach, Florida
  - University of Miami, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - NanoHealth Associates, Miami Beach, Florida
  - Urology Center of Florida, Pompano Beach, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Investigative Clinical Research of Indiana, Elwood, Indiana
  - Urology of Indiana, Indianapolis, Indiana
  - Tandem Clinical Research GI, LLC, Marrero, Louisiana
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Premier Urology Group, Edison, New Jersey
  - ProHEALTH Care Associates, Garden City, New York
  - AccuMed Research Associates, Garden City, New York
  - NYU Langone Health, New York, New York
  - The Research Foundation for the State University of New York at Buffalo, Williamsville, New York
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Warren Alpert School of Medicine Brown University, Providence, Rhode Island
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - North Austin Urology, Austin, Texas
  - Coastal Bend Clinical Research, Corpus Christi, Texas
  - Prime Revival Research Institute, Flower Mound, Texas
  - Baylor College of Medicine, Houston, Texas
  - Crossroads Clinical Research, Victoria, Texas

IPD SHARING:
Plan to Share IPD: No